CLINICAL TRIAL: NCT06055140
Title: Evaluation of Thoracolumbar Fascia and Relationship With Low Back Pain in Individuals With Idiopathic Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gözde Yagci (Gür), Associate Professor, Hacettepe University
Other Study IDs: GO 23/516
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Idiopathic Scoliosis; Pain
Keywords: fascia; scoliosis; pain
MeSH Terms: conditions — Pain; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Idiopathic scoliosis without pain: In this group, there will be individuals diagnosed with idiopathic scoliosis whose Cobb angle is above 15 degrees and whose pain level, as assessed by the Visual Analog Scale, is below 3.
- Idiopathic scoliosis with pain: In this group, there will be individuals diagnosed with idiopathic scoliosis whose Cobb angle is above 15 degrees, and their pain level, as assessed by the Visual Analog Scale, is above 3.
- Control: In this group, there will be healthy individuals whose pain level, as assessed by the Visual Analog Scale, is below 3.

SUMMARY:
This observational study seeks to explore the potential association between thoracolumbar fascia characteristics and low back pain in individuals diagnosed with idiopathic scoliosis.

DETAILED DESCRIPTION:
This observational study aims to investigate the potential link between thoracolumbar fascia characteristics and low back pain in individuals with idiopathic scoliosis. The hypothesis underlying this study posits that alterations in thoracolumbar fascia thickness and properties contribute to changes in trunk flexibility and subsequently influence the occurrence and intensity of low back pain in patients with idiopathic scoliosis. The researchers believe that an increase in thoracolumbar fascia thickness may lead to reduced trunk flexibility, restricting the normal range of motion and potentially causing or exacerbating low back pain.

To explore this hypothesis, the study will include participants diagnosed with idiopathic scoliosis. The researchers will measure thoracolumbar fascia thickness using ultrasound and assess trunk flexibility through various range of motion tests, including trunk flexion, extension, and lateral flexion using a goniometer, as well as the sit-and-reach test. To quantify the severity of the spinal curvature, the Cobb angle will be measured on anteroposterior standing radiographs.

Participants will also be asked to report their pain levels using the Visual Analog Scale, a simple tool where individuals rate their pain on a scale from 0 to 10. By analyzing the collected data, the researchers aim to establish potential correlations between thoracolumbar fascia thickness, trunk flexibility, and low back pain in individuals with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria (with Scoliosis):

1. Being 10 years of age or older
2. Having a diagnosis of idiopathic scoliosis
3. Having a Cobb angle measurement above 15 degrees

Inclusion Criteria (for Healthy Individuals):

1. Being 10 years of age or older
2. Have no pathological spinal curvature.
3. Have no history of low back pain in the last 3 months (Visual Analog Scale score <3/10).

Exclusion Criteria:

1. Having any neurological, psychological, congenital, or rheumatological condition
2. Having a history of surgery or trauma involving the lower extremities or spinal region within the last 1 year
3. Having received any previous treatment related to scoliosis

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected using snowball sampling from individuals diagnosed with idiopathic scoliosis and aged 10 years or older, who meet the inclusion criteria. Snowball sampling involves initially recruiting participants who meet the inclusion criteria and then asking them to refer other potential participants from their social network who also have idiopathic scoliosis. Exclusion criteria will involve individuals with neurological, psychological, congenital, or rheumatological conditions, those with a history of surgery or trauma involving the lower extremities or spinal region within the last 1 year, and individuals who have received any previous treatment related to scoliosis.
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Thoracolumbar Fascia Thickness | Baseline
  The thoracolumbar fascia thickness (mm) obtained after ultrasonographic assessment.

SECONDARY OUTCOMES:
Visual analog scale | Baseline
  The pain levels of individuals obtained after the Visual Analog Scale assessment.Patients will be asked to mark their perceived pain levels on a 100-millimeter horizontal line.
Trunk Normal Range of Motion | Baseline
  The degrees of trunk flexion, extension, right lateral flexion, and left lateral flexion obtained after goniometric measurements.
Trunk Flexibility | Baseline
  The sit-and-reach test and trunk rotation values will be recorded in centimeters.
McGill Short Form Pain Questionnaire | Baseline
  A questionnaire providing numerical outputs about the sensory qualities, affective qualities, and intensity of pain.
Oswestry Low Back Pain Disability Questionnaire | Baseline
  A questionnaire scored from 0 to 50, assessing the impact of low back pain on daily life activities.
Scoliosis Research Society-30 (SRS-30) | Baseline
  This questionnaire consists of 30 questions and is used to evaluate the health-related quality of life in individuals with scoliosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Yerli, MSc, PT, Principal Investigator — Hacettepe University; Satuk Bugrahan Yinanc, MSc, PT, Principal Investigator — Hacettepe University; Gözde Yağcı, PhD, PT, Study Director — Hacettepe University; Fatih Erbahçeci, PhD, PT, Study Director — Hacettepe University; Levent Özçakar, Phd, MD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Institute of Health Sciences, Faculty of Physical Therapy and Rehabilitation, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choudhry MN, Ahmad Z, Verma R. Adolescent Idiopathic Scoliosis. Open Orthop J. 2016 May 30;10:143-54. doi: 10.2174/1874325001610010143. eCollection 2016. PMID 27347243
- [Background] Pirri C, Pirri N, Guidolin D, Macchi V, Porzionato A, De Caro R, Stecco C. Ultrasound Imaging of Thoracolumbar Fascia Thickness: Chronic Non-Specific Lower Back Pain versus Healthy Subjects; A Sign of a "Frozen Back"? Diagnostics (Basel). 2023 Apr 16;13(8):1436. doi: 10.3390/diagnostics13081436. PMID 37189537